CLINICAL TRIAL: NCT03635021
Title: Phase III Randomized Sequential Open-label Study to Evaluate the Efficacy of FOLFOX + Panitumumab Followed by FOLFIRI + Bevacizumab (Sequence 1) Versus FOLFOX + Bevacizumab Followed by FOLFIRI + Panitumumab (Sequence 2) in Untreated Patients With Wild-type RAS Metastatic, Primary Left-sided, Unresectable Colorectal Cancer: The CR-SEQUENCE
Brief Title: Study to Evaluate the Efficacy of FOLFOX + Panitumumab Followed by FOLFIRI + Bevacizumab (Sequence 1) Versus FOLFOX + Bevacizumab Followed by FOLFIRI + Panitumumab (Sequence 2) in Untreated Patients With Wild-type RAS Metastatic, Primary Left-sided, Unresectable Colorectal Cancer
Acronym: CR-SEQUENCE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-18-01
Record Dates: First submitted 2018-08-09; First posted 2018-08-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; FOLFOX; FOLFIRI; panitumumab; bevacizumab; wild-type RAS; primary left-sided
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Panitumumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): FOLFOX regimen panitumumab FOLFIRI regimen bevacizumab
  Interventions: Drug: FOLFOX regimen; Drug: Panitumumab; Drug: Bevacizumab; Drug: FOLFIRI regimen
- Sequence 2 (Experimental): FOLFOX regimen bevacizumab FOLFIRI regimen panitumumab
  Interventions: Drug: FOLFOX regimen; Drug: Panitumumab; Drug: Bevacizumab; Drug: FOLFIRI regimen

INTERVENTIONS:
Drug: FOLFOX regimen — oxaliplatin 85 mg/m2 administered by IV infusion over 120 minutes on Day 1, L-leucovorin 200 mg/m2 administered as a 2-hour IV infusion on Day 1 and 5-FU 400 mg/m2 administered as IV bolus over approximately 2 to 4 minutes on Day 1 followed by 5-FU 2400 mg/m2 administered as IV infusion over 46- 48 hours on Days 1 and 2
Drug: Panitumumab — 6 mg/kg administered by intravenous (IV) infusion over 60 minutes on Day 1 of each 14-day cycle
Drug: Bevacizumab — 5 mg/kg administered by IV infusion over 60 minutes on Day 1 of each 14-day cycle
Drug: FOLFIRI regimen — irinotecan 180 mg/m2 administered as a 90 minutes IV infusion on Day 1, L-leucovorin 200 mg/m2 administered as a 2-hour IV infusion on Day 1 and 5-FU 400 mg/m2 administered as IV bolus over approximately 2 to 4 minutes on Day 1 followed by 5-FU 2400 mg/m2 administered as IV infusion over 46-48 hours on Days 1 and 2

SUMMARY:
The purpose of this study is to assess the efficacy of FOLFOX + panitumumab followed by FOLFIRI + bevacizumab (Sequence 1) versus FOLFOX + bevacizumab followed by FOLFIRI + panitumumab (Sequence 2) in untreated patients with wild-type RAS metastatic, primary left-sided, unresectable colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman at least 18 years old.
2. Capable of understand, sign and date an informed consent approved by an IEC.
3. Histologically confirmed adenocarcinoma of the left colon or rectum (originate in the splenic flexure, descending colon, sigmoid colon, or rectum) in patients with unresectable (not amenable to radical surgery of metastases at the study inclusion) metastatic (M1) disease.
4. Patients who had wild-type RAS status confirmed as per standard of care according to international guidelines prior to first-line initiation.

   *RAS analysis should include at least KRAS exons 2, 3 and 4 (codons 12, 13, 59, 61, 117 and 146) and NRAS exons 2, 3 and 4 (codons 12, 13, 59, 61 and 117)
5. At least one unidimensionally measurable lesion per RECIST criteria (version 1.1).
6. ECOG performance status < 2.
7. Adequate bone marrow function: neutrophils ≥1.5 x109 / L; platelets ≥100 x109 /L; haemoglobin ≥ 9 g/dL.
8. Hepatic, renal and metabolic function as follows:

   * Total bilirubin count ≤1.5 x upper limit of normal (ULN), serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) and serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) ≤ 2.5 x ULN (5 x ULN for subjects with liver involvement of their cancer or 10 x ULN for subjects with bone involvement).
   * Renal function, calculated as creatinine clearance or 24-hour creatinine clearance ≥ 50 mL/min.

Exclusion Criteria:

1. History of prior or concurrent central nervous system metastases.
2. History of another primary cancer, except: curatively treated in situ cervical cancer, or curatively resected non-melanoma skin cancer, or other primary solid tumour curatively treated with no known active disease present and no treatment administered for ≥ 5 years before randomization.
3. Prior chemotherapy or other systemic anticancer therapy for treatment of metastatic colorectal carcinoma.
4. Prior adjuvant chemotherapy for colorectal cancer (stage I, II or III) terminated less than 6 month before metastatic disease was diagnosed.
5. Unresolved toxicities of a previous systemic treatment that, in the opinion of the Investigator, cause the patient unfit for inclusion.
6. Prior use (as monotherapy or adjuvant treatment) of anti-EGFR antibody therapy (e.g. cetuximab), anti-VEGF or small molecule EGFR inhibitors (e.g. erlotinib).
7. Prior hormonal therapy, immunotherapy or approved or experimental antibody/proteins ≤ 30 days before inclusion.
8. Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiating study treatment or a history of ventricular arrhythmia.
9. Uncontrolled hypertension.
10. History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest computerised tomography (CT).
11. Treatment for systemic infection within 14 days before the start of study treatment.
12. Acute or subacute intestinal occlusion and/or active inflammatory bowel disease or other bowel disease that causes chronic diarrhoea (defined as grade ≥ 2 diarrhoea according to NCI-CTCAE version 4.03).
13. Clinically significant peripheral sensory neuropathy.
14. Evidence of previous acute hypersensitivity reaction, of any grade, to any component of the treatment.
15. History of Gilbert disease or known dihydropyrimidine deficiency syndrome.
16. Recent (within 6 months before the start of study treatment) gastroduodenal ulcer to be active or uncontrolled.
17. Recent (within 6 months before the start of study treatment) pulmonary embolism, deep vein thrombosis, or other significant venous event.
18. Pre-existing bleeding diathesis and/or coagulopathy with exception of well-controlled anticoagulation therapy (within 6 months before the start of study treatment)
19. Recent (within 4 weeks prior to inclusion in the study) major surgical procedure, open biopsy, or significant traumatic injury not yet recovered from prior major surgery
20. History of any disease that may increase the risks associated with study participation or may interfere with the interpretation of study results.
21. Known positive test for human immunodeficiency virus infection, hepatitis C virus, and chronic active hepatitis B infection.
22. Any disorder that compromises the patient's ability to provide written informed consent and/or comply with study procedures.
23. Any investigational agent within 30 days prior to inclusion.
24. Pregnant or breastfeeding woman.
25. Surgery (excluding diagnostic biopsy or placement of a central venous catheter) and/or radiotherapy within 28 days prior to inclusion in the study.
26. Male or female of childbearing age who do not agree with taking adequate contraceptive precautions, i.e. use contraception double barrier (e.g. diaphragm plus condoms) or abstinence during the course of the study and for 6 months after the last administration of study drug for women and 1 month for men.
27. The patient is unwilling or unable to meet the requirements of the study.
28. Psychological, geographical, familial or sociological conditions that potentially prevent compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate at 35 months | 35 months after date of randomization
  35-month PFSR defined as the number of patients, who at 35 months after randomization, have not had second or first disease progression nor died (due to any cause), over the total number of evaluable patients.

SECONDARY OUTCOMES:
overall survival rate at 35 months | 35 months after date of randomization
  35-month OSR defined as the number of patients who at 35 months after randomization have not died over the total number of evaluable patients.
overall survival | Baseline through the end of the study (up 72 months)
  OS defined as the time from randomization to the date of death (due to any cause), with patients alive or lost to follow-up at the analysis data cut-off date censored at their last contact date.
progression-free from randomization to second progression or death | Baseline through the end of the study (up 72 months)
  Total PFS defined as the time from randomization to second disease progression (i.e. progression during the second-line treatment) or death (due to any cause).
progression-free survival in first-line treatment and in second-line treatment | Baseline through the end of the study (up 72 months)
  PFS in first-line treatment defined as the time from randomization to disease progression or death (due to any cause) during first-line treatment. PFS in second-line treatment defined as the time from the date of second-line treatment initiation to disease progression or death (due to any cause) during secondline treatment.
time to first-line treatment failure and to second-line treatment failure | 72 months
  Time to first-line treatment failure defined as the time form randomization to disease progression, death (due to any cause) or discontinuation due to toxicity during first-line treatment. Time to second-line treatment failure defined as the time from the date of second-line treatment initiation to disease progression, death (due to any cause) or discontinuation due to toxicity during second-line treatment.
objective response rate | Baseline through the end of the study (up 72 months)
  Proportion of patients with an objective response (complete or partial response) per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria in first-line treatment and in second-line treatment.
proportion of patients with Early Tumour Shrinkage | Baseline through the end of the study (up 72 months)
  Proportion of patients with ETS in first-line treatment and in second-line treatment. ETS will be defined as a reduction in tumour size ≥30% (RECIST 1.1 criteria) at the first evaluation (i.e. week 12)
Depth of Response | Baseline through the end of the study (up 72 months)
  DpR measured as the maximum decrease in target measurement (RECIST 1.1 criteria) during the complete course of evaluation in first-line treatment and in second-line treatment.
disease control rate | Baseline through the end of the study (up 72 months)
  Proportion of patients with disease control (complete, partial response or stable disease) in first-line treatment and in second-line treatment.
duration of disease control | Baseline through the end of the study (up 72 months)
  Duration of disease control defined as time from first confirmed disease control to disease progression per RECIST 1.1 criteria or death (due to any cause) in first-line treatment and in second-line treatment. For patients with disease control who have not progressed or died at last observation, duration of disease control will be censored at their last evaluable disease assessment date.
duration of response | Baseline through the end of the study (up 72 months)
  Duration of response defined as time from first confirmed objective response to disease progression per RECIST 1.1 criteria or death (due to any cause) in first-line treatment and in second-line treatment. For patients with response who have not progressed or died at last observation, duration of response will be censored at their last evaluable disease assessment date.
time to response | Baseline through the end of the study (up 72 months)
  Time to response in first-line treatment defined as the time from randomization to the date of first confirmed objective response per RECIST 1.1 criteria during first-line treatment.
  Time to response in second-line treatment defined as the time from the date of second-line treatment initiation to the date of first confirmed objective response per RECIST 1.1 criteria during second-line treatment.
Incidence and severity of AEs CTCAE v4.03 criteria | Baseline through the end of the study (up 72 months)
  Safety assessment will consist of monitoring adverse events (AEs), including AEs of special interest, serious AEs (SAEs) and laboratory safety parameters. AEs will be graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03.

OTHER OUTCOMES:
Impact of baseline biomarkers predictive of the efficacy | Baseline through the end of the study (up 72 months)
  Efficacy variables according different baseline biomarkers.
clinical impact of clonal dynamics by longitudinal analysis of circulating tumour deoxyribonucleic acid (ctDNA) in plasma | Baseline through the end of the study (up 72 months)
  Proportion of patients with emerging mutations of resistance to targeted therapies. Blood samples at various timepoints and tumour tissue sample will be collected in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Salazar, MD, PhD, Study Chair — Instituto Catalán de Oncología. Hospital Duran i Reynals; Alfredo Carrato, MD, PhD, Study Chair — Hospital Universitario Ramon y Cajal
Locations (1):
- Spanish Cooperative Group for the Treatment of Digestive Tumors, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No